CLINICAL TRIAL: NCT04419181
Title: A Feasibility Study of De-escalation of Chemotherapy in Patients With Early-Stage HER2 Positive Breast Cancer
Brief Title: Feasibility of Chemotherapy De-escalation in Early-Stage HER2 Positive Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in the landscape of current treatment of early stage breast cancer. Larger clinical trials answering similar questions are expected to result in the next few years.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Ajay Dhakal, Assistant Professor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBRS20013
Record Dates: First submitted 2020-06-01; First posted 2020-06-05 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: HER2-positive Breast Cancer
Keywords: HER2-positive Breast Cancer; De-escalation
MeSH Terms: interventions — Docetaxel; Carboplatin; Trastuzumab; pertuzumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to an arm of the trial based on their outcomes after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pathologic complete response (pCR) (Experimental): Participants will receive four cycles of TCHP [docetaxel (Taxotere®), carboplatin, trastuzumab (Herceptin®), pertuzumab], followed by surgery. Participants who achieve pathologic complete response will receive infusions of trastuzumab every 3 weeks for a total of 12 cycles/infusions.
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab
- Residual Disease (Experimental): Participants will receive four cycles of TCHP [docetaxel (Taxotere®, carboplatin, trastuzumab (Herceptin®), pertuzumab], followed by surgery. Participants who have residual disease may be offered two more cycles of TCHP in the adjuvant settings (optional) per treating oncologist's discretion and then will receive infusion of Trastuzumab Emtansine (TDM1) plus pertuzumab every three weeks for a total of 12 cycles/infusions.
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: Docetaxel — Dose: 75 mg/m2 q3w
  Other Names: Taxotere
Drug: Carboplatin — Dose: area under the concentration-time curve [AUC] 6 q3w
  Other Names: Paraplatin
Drug: Trastuzumab — Dose: 8-mg/kg loading dose, 6-mg/kg maintenance dose q3w
  Other Names: Herceptin
Drug: Pertuzumab — Dose: 840-mg loading dose, 420-mg maintenance dose q3w
  Other Names: Perjeta
Drug: Trastuzumab emtansine — Dose: 3.6mg/kg q3w
  Other Names: TDM1
  Arms: Residual Disease

SUMMARY:
The main purpose of this research study is to find out if de-escalation of chemotherapy before surgery followed by a selective escalation of adjuvant targeted therapies are efficacious and tolerable in early-stage HER2 positive breast cancer.

DETAILED DESCRIPTION:
Assess the feasibility of four cycles of neoadjuvant Docetaxel Carboplatin Trastuzumab and Pertuzumab (TCHP) in women with early-stage (local/locally advanced) HER2+ breast cancer with a selective escalation of targeted HER2 directed therapy in the high risk group in the adjuvant setting. Participants with any residual disease after four cycles of TCHP will receive Trastuzumab Emtansine (TDM1) plus Pertuzumab while those with complete pathological response will receive Trastuzumab in the adjuvant settings.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years of age
* Biopsy proven HER2+ early breast cancer
* ECOG performance status 0-1
* Should be a candidate for neoadjuvant chemotherapy using standard guidelines of tumor size of 2cm or more and /or axillary lymph node-positive disease.
* Adequate cardiac, bone marrow, kidney, and liver functions per treating physician's discretion.
* Women of childbearing potential who are sexually active must agree to use highly effective methods of contraception during treatment and for three weeks after the last dose of chemotherapy or anti-HER2 therapy. The women currently using hormonal contraceptives must agree to change to an alternative highly effective method of contraception
* Willingness and ability to comply with study and follow-up procedures and give written informed consent.

Exclusion Criteria:

* Any evidence of stage IV breast cancer
* Participant deemed unsuitable for clinical trial enrolment by treating physician based on the participants' compliance, location and commute requirements, or tolerance of therapies involved
* Any invasive malignancy within the last two years of study enrollment except for adequately treated basal cell carcinoma, squamous cell carcinoma, or non-melanoma skin cancer.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
One Year Invasive Disease-Free Survival | One year from the breast cancer surgery
  The study will be considered feasible if the researchers observe the invasive disease free survival (IDFS) estimate at one year to be 90% or more among those who achieved a pCR, or if the researchers observe the IDFS estimate at one year to be 85% or more among those who had residual disease.

SECONDARY OUTCOMES:
Pathologic Complete Response rate | 12 weeks from start of treatment
  Assess the pCR rate after four cycles (12 weeks) of TCHP.
Toxicity of chemo and HER2 therapies | One year from the start of treatment
  Evaluate toxicity associated with neoadjuvant and adjuvant chemo and/or HER2 directed therapies. Percentage of grade 1 to grade 5 toxicities will be assessed during the neo-adjuvant TCHP therapy for all participants. Percentage of grade 1 to grade 5 toxicities will be assessed with adjuvant trastuzumab therapy for the cohort with pathological complete response, and with optional adjuvant TCHP therapy and adjuvant TDM1 + pertuzumab therapy for the residual disease cohort. Toxicity data will be obtained based on the clinical assessment of the participants by the investigators and based on laboratory data.
Two Year Invasive Disease-Free Survival | Two years from the breast cancer surgery
  Two year invasive disease-free survival (IDFS) of participants with pCR and participants with residual disease

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Dhakal, MBBS, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States